CLINICAL TRIAL: NCT03989401
Title: If Muti-media Health Education Reduces the Workload of Nurses Without Affecting Patient's Satisfaction:a Perspective Randomized Controlled Trial
Brief Title: Effect of Multi-media Health Education on Nurses' Workload and Patient's Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Jia Yao, Ph.D Clinical research administration officer, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Multi-media health education
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Health Education
Keywords: Nurse; Workload; Multimedia; Patients Satisfaction; Surgery; Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimedia video education (Experimental): The experimental group conducted multimedia video education while admission.
  Interventions: Other: Multimedia video health education
- None multimedia video education (No Intervention): The control group conducted usual nursing of oral face-to-face education on admission.

INTERVENTIONS:
Other: Multimedia video health education — The experimental group conducted multimedia video education while admission.
  Arms: Multimedia video education

SUMMARY:
Assessing whether multi-media health education reduce nurse workload and does not decrease the satisfaction of patients in surgical ward when admission.

DETAILED DESCRIPTION:
Operation usually causes severe physical and mental stress to the patients, mainly because of fear and anxiety caused by patients worrying about the uncertainty about surgery, and finally affecting the patient's surgical efficacy and recovery. This is the main reason in terms of surgical nurse workload is much more than those internal medicine nurse.

As a major part of nursing work, health education has especially important to patients. The quality and efficiency of health education directly affects the rehabilitation of patients. It can help patients correctly understand the relevant knowledge of disease and master the skills of recovery.

At present, the health education in surgery department is mainly carried out by oral face-to-face communication and guidance from admission nurses. This kind of education method showed time-consuming and laborious.In addition, oral guidance is more reliable on nurse ability of expression and acknowledgement. Multimedia-based health education is an update mode combined with audio-visual stimulation and patients' own participation. Mobile terminal makes patient more acceptable, flexible, standardized in receiving the health education during hospitalization. This prospective study is aimed to assess whether multimedia-video education could reduce nurse workload and do not decrease the satisfaction of surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with general diseases and who need surgical treatment
* Primary school or above education history, with clear awareness, can cooperate with the collection of clinical data, and can communicate in Chinese
* Patients who signed the informed consent

Exclusion Criteria:

* Patients with visual and hearing impairment
* Patients with mental illness, dementia and other mental disorders
* Patients with complications of heart, brain and nephropathy
* Patients who cannot take care of themselves
* Emergency and critically ill patients
* Patients participated other research

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Nursing workload | 1 month
  Daily working hours for admission nurses on patients guidance on the first 24 hours in hospital, include the length of guidance time and the inquiry times.
The satisfaction of patients, family members, doctors and nurses about health education: Questionnaire | 1 month
  The questionnaires were designed by ourselves according to relevant research and literature, to quantify the level of satisfaction on admission health education for patients and family members, and also doctors and nurses .
  The patients and family members satisfaction questionnaire has 11 satisfaction questions, which scored on a scale of 1-5(one to five stars, one star represents unsatisfactory, five stars represent highly satisfactory). The scores range from 11-55.
  * 11-21 Unsatisfactory
  * 22-32 Not quite satisfactory
  * 33-43 Generally satisfactory
  * 44-55 Highly satisfactory
  The doctors and nurses satisfaction questionnaire has 15 satisfaction questions, which scored on a scale of 1-5(one to five stars, one star represents unsatisfactory, five stars represent highly satisfactory). The scores range from 15-75.
  * 15-29 Unsatisfactory
  * 30-44 Not quite satisfactory
  * 45-59 Generally satisfactory
  * 60-75 Highly satisfactory

SECONDARY OUTCOMES:
Patients' anxiety level before and after health education: Zung Self Rating Anxiety Scale（SAS） | 1 month
  The Zung Self-Rating Anxiety Scale (SAS) is an anxiety measure designed by William WK Zung to quantify the level of anxiety for patients experiencing anxiety related symptoms.
  The self-administered test has 20 questions. Each question is scored on a scale of 1-4 (none or a little of the time, some of the time, good part of the time, most of the time). There are fifteen questions worded toward increasing anxiety levels and five questions worded toward decreasing anxiety levels.
  The scores range from 20-80.
  * 20-44 Normal Range
  * 45-59 Mild to Moderate Anxiety Levels
  * 60-74 Marked to Severe Anxiety Levels
  * 75-80 Extreme Anxiety Levels
Inquiry times on health education content of patients family members | 1 month
  The exactly times of patient's family members ask nursing staff for health education content.
The times of patients and their family members watched the health education videos | 1 month
  The times of patients and their family members watched the health education videos.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Yao, Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Jia Yao, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacob C, Sanchez-Vazquez A, Ivory C. Clinicians' Role in the Adoption of an Oncology Decision Support App in Europe and Its Implications for Organizational Practices: Qualitative Case Study. JMIR Mhealth Uhealth. 2019 May 3;7(5):e13555. doi: 10.2196/13555. PMID 31066710
- [Result] Hindi AMK, Seston EM, Bell D, Steinke D, Willis S, Schafheutle EI. Independent prescribing in primary care: A survey of patients', prescribers' and colleagues' perceptions and experiences. Health Soc Care Community. 2019 Jul;27(4):e459-e470. doi: 10.1111/hsc.12746. Epub 2019 Mar 18. PMID 30884013
- [Derived] Yang L, Qin Z, Yao J, Xu H, Tian J, Ren Y, Wang H, Meng W. Enhancing patient satisfaction and reducing nurse workload: the impact of multimedia health education in a prospective single-center randomized controlled trial. Front Med (Lausanne). 2025 Feb 19;12:1400061. doi: 10.3389/fmed.2025.1400061. eCollection 2025. PMID 40046935